CLINICAL TRIAL: NCT01319786
Title: Effect of a Polyphenol Rich Diet on Vascular and Platelet Function- a Randomised Control Trial
Brief Title: Effect of a Polyphenol Rich Diet on Vascular and Platelet Function
Acronym: PPhIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Rebecca Noad, Professor Pascal McKeown, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QueensUBelfast
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
Keywords: Hypertension; Microvascular function
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low- polyphenol diet (Other)
  Interventions: Other: Two portions of fruit and vegetables per day (excluding berries and dark chocolate)
- High-polyphenol diet (Active Comparator)
  Interventions: Other: Six portions of fruit and vegetables per day (one of which must be berries) and 50g dark chocolate.

INTERVENTIONS:
Other: Two portions of fruit and vegetables per day (excluding berries and dark chocolate) — Two portions of fruit and vegetables per day (excluding berries and dark chocolate)
  Arms: Low- polyphenol diet
Other: Six portions of fruit and vegetables per day (one of which must be berries) and 50g dark chocolate. — Six portions of fruit and vegetables per day (one of which must be berries) and 50g dark chocolate.
  Arms: High-polyphenol diet

SUMMARY:
Previous work has shown that increasing fruit and vegetable intake in patients with high blood pressure improves cardiovascular function. Research indicates that this may be partly owing to compounds called polyphenols, which are found in abundance in fruits and vegetables and other foods such as wine, tea and dark chocolate. The investigators now wish to test if consuming fruits and vegetables (including berries which are very rich in polyphenols), as well as dark chocolate, has further benefits for cardiovascular function. A total of 110 subjects with high blood pressure will be recruited and asked to follow a low polyphenol diet (2 portions of fruit and vegetables daily and no berries or dark chocolate) for four weeks (a washout period). They will then be randomised to continue this diet or to consume 6 portions of fruits and vegetables (to include 1 portion berries) and 1 portion of dark chocolate daily for 8 weeks. The fruit, vegetables and dark chocolate will be provided free of charge and delivered to the homes of the participants who are randomised to the high fruit and vegetable arm of the study.

Assessment of microvascular and platelet function will be undertaken before and after consuming this diet. Improvements in these tests of cardiovascular function have previously been linked to reduced risks of heart disease in people with high blood pressure. This study will provide evidence as to whether or not a polyphenol rich diet can reduce the risk of developing heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65 years old
* Systolic blood pressure 140-179 mmHg or diastolic blood pressure 90-109 mmHg

Exclusion Criteria:

* diabetes mellitus
* an acute coronary syndrome or transient ischaemic attack within the past 3 months
* special dietary requirements, food sensitivities or vegetarian/vegan diet by choice
* oral anticoagulation therapy
* body mass index greater than 35kg/m2
* excessive alcohol consumption (defined as > 28 units/week in men and 21 units/week in women)
* fasting triglyceride concentration > 4 mmol/l
* pregnancy/lactation
* taking antioxidant supplements
* medical conditions or dietary restrictions that would substantially limit ability to complete the study requirements

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Vascular function | Measured at weeks 4 and 12
  Pharmacological provocation of endothelium-dependent vasomotion.

SECONDARY OUTCOMES:
Platelet function, biomarkers of cardiovascular risk and heart rate variability | Measured at weeks 0, 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Pascal McKeown, MD, Principal Investigator — Belfast Health and Social Care Trust; Jayne Woodside, PhD, Study Director — Queen's University, Belfast; Michelle McKinley, PhD, Study Director — Queen's University, Belfast
Locations (1):
- Belfast Health and Social Care Trust, Belfast, United Kingdom

REFERENCES:
- [Derived] Noad RL, Rooney C, McCall D, Young IS, McCance D, McKinley MC, Woodside JV, McKeown PP. Beneficial effect of a polyphenol-rich diet on cardiovascular risk: a randomised control trial. Heart. 2016 Sep 1;102(17):1371-9. doi: 10.1136/heartjnl-2015-309218. Epub 2016 May 10. PMID 27164919